CLINICAL TRIAL: NCT06694363
Title: New Biomarker-based Strategy to Screen and Monitor for Activated Phosphoinositide 3-kinase Δ Syndrome
Acronym: BIO-APDS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240329; 2024-A01816-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Activated PI3K Delta Syndrome
Keywords: Activated PI3K delta syndromes; APDS; Leniolisib
MeSH Terms: conditions — Activated PI3K-delta Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1 - initiating treatment: 10 patients with a genetic diagnosis of APDS type 1 or type 2 who are to be treated with a selective PI3Kδ inhibitor, Lenolisib.
  Interventions: Biological: Blood samples; Biological: Urine samples; Biological: Stool samples
- 2 - already on treatment: 4 patients with a genetic diagnosis of APDS type 1 or type 2 already treated with a selective PI3Kδ inhibitor, Lenolisib.
  Interventions: Biological: Blood samples; Biological: Urine samples; Biological: Stool samples

INTERVENTIONS:
Biological: Blood samples — A maximum of 27 ml of blood collected at each visit for metabolic markers analysis
Biological: Urine samples — One urine sample collected at each visit for enteric virus infection research
Biological: Stool samples — One stool sample collected at each visit for enteric virus infection research

SUMMARY:
The study would like to compare patient samples at different time points using state-of the art-phenotyping tools.

Collection of blood samples of APDS patients undergoing PI3K inhibitor treatment will be collected when feasible according to the standard of care planning (a blood test is supposed to be performed for these patients at M0-M3-M6-M12 then each 6 months for a total period of 2 years from the beginning of the PI3K inhibitor treatment).

The whole blood will be processed in order to isolate the peripheral blood mononuclear cells (PBMC) and the plasma. Serum, RNA and DNA extraction will be performed on a separate sample.

DETAILED DESCRIPTION:
Activated PI3K delta syndromes (PI3Kδ) (APDS type 1 and type 2) are combined immunodeficiencies with variable clinical manifestations caused by heterozygous gain-of-function mutations of the PIK3CD gene. APDS is a very young onset disease, most clinical manifestations appear in pediatric age. Patients may experience severe, disabling, and life-threatening clinical manifestations. Additionally, they may exhibit autoimmunity in addition to immune deficiency. APDS patients present a high risk of developing tumors especially B lymphomas. Hematopoietic stem cell transplantation (HSCT) is the only curative option and, given the risks, may be considered for patients with severe APDS (including those who have developed lymphoma). HSCT is curative, but carries a 10 to 20% mortality risk and cannot guarantee reversibility of organ damage. Positive data from the phase II/III study of the PI3Kδ selective inhibitor leniolisib met the co-primary criteria of reduced lymph node size and increased percentage of B naïve cells in patients with APDS. In addition, safety data from the study showed that leniolisib was well tolerated by participants. The drug is also under review by the European Medicines Agency and a marketing authorization for APDS patients older than 12 years old will be soon available. In the meantime the access to this drug is available by compassionate use for patients older than 12 years old.

In this context, it will be interesting to evaluate the clinical and biological profile of these patients before and after leniolisib treatment in order to identify useful biomarkers for the follow up of the disease. In addition, carful long-term monitoring of patients under PI3Kδ inhibitors is mandatory to detect adverse effects of iatrogenic overinhibition of the PI3K pathway.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Patients with genetic diagnosis of APDS type 1 or type 2 and planned to be treated by PI3Kδ selective inhibitor leniolisib
* Primary immunodeficient patients with new disease-causing variants in the PIK3CD gene or PIK3R1 gene
* Minimum age 12 years old
* Patients or holders of parental authority do not oppose participation in this research.
* Patients affiliated to a Health Insurance scheme or beneficiaries

Group 2 :

* Patients with genetic diagnosis of APDS type 1 or type 2 already treated by PI3Kδ selective inhibitor leniolisib in the last 2 years
* Patients whose pre-treatment samples are available/analyzable
* Minimum age 12 years old
* Patients or holders of parental authority do not oppose participation in this research.
* patients affiliated to a Health Insurance scheme or beneficiaries

Exclusion Criteria:

* Bone marrow transplantation
* Refusal to participate to the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetic diagnosis of APDS type 1 or type 2 and planned to be treated by PI3Kδ selective inhibitor leniolisib and patients with genetic diagnosis of APDS type 1 or type 2 already treated by PI3Kδ selective inhibitor leniolisib in the last 2 years
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Biomarker | At 0 day, 3 months, 6 months, 12 months, 18 months and 24 months of treatment
  Identify new biomarker marker for increased PI3K signaling to monitor the disease severity by mass cytometry, single cell RNA-sequencing, single cell ATAC-sequencing and screening for auto-antibodies

SECONDARY OUTCOMES:
activation-induced cytidine deaminase (AID) off-target activity | At 0 day, 3 months, 6 months, 12 months, 18 months and 24 months of treatment
  Investigate the possibility of activation-induced cytidine deaminase (AID) off-target activity in memory B cells due to PI3Kdelta inhibitor treatment by NGS panel sequencing
Correlation between biological data with the clinical data | At 0 day, 3 months, 6 months, 12 months, 18 months and 24 months of treatment
  the analyses results will be correlated with the clinical data collected for the patients enrolled in the trial and receiving PIK3CD inhibitor treatment (early access program) in order to explore a possible correlation between biological data and clinical characteristics.
Enteric virus infection research | At 0 day, 3 months, 6 months, 12 months, 18 months and 24 months of treatment
  Presence of Chronic enteric virus infection will be investigated by multiplex PCR and if negative by NGS in stools, plasma, urins

CONTACTS AND LOCATIONS:
Overall Officials: Sven Kracker, PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (7):
- France (7):
  - Hôpital Haut Levêque - BORDEAUX, Bordeaux
  - Hôpital Pellerin Enfants - BORDEAUX, Bordeaux
  - Hôpital Jeanne de Flandres - LILLE, Lille
  - Hôpital La Timone adulte - MARSEILLE, Marseille
  - Hôpital Necker Enfants Malades - PARIS, Paris
  - CHU IUCT Oncopole - TOULOUSE, Toulouse
  - Hôpital des enfants - TOULOUSE, Toulouse

IPD SHARING:
Plan to Share IPD: No